CLINICAL TRIAL: NCT02980835
Title: Optimal Timing of Intercostal Nerve Blocks During Video-Assisted Thoracic Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: The VA Western New York Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nader D Nader, Professor and Senior Vice Chair, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 721921
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Video-Assisted Thoracic Surgery; Video-Assisted Thoracoscopic Surgery
MeSH Terms: interventions — Saline Solution; Ropivacaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Patients who receive injections of A (a total of a 10 mL-solution that consists of 9 mL of ropivacaine HCl 0.5% and 1 mL of dexamethasone 4mg/mL preparation) at the beginning of surgery and second set of injections containing a mixture of B (contains 10 mL of 0.9% normal saline) and C (a total 25 mL solution that consists of 24 mL of ropivacaine HCl 0.5%, 1 mL of dexamethasone-4mg/mL preparation, and 0.125 mL of epinephrine-1:1000 preparation) prior to the closure
  Interventions: Drug: Normal Saline; Drug: Ropivacaine; Drug: Epinephrine; Drug: Dexamethasone
- Control (Active Comparator): Participants who receive injection of B (contains 10 mL of 0.9% normal saline) at the beginning of surgery and injectate A (a total of a 10 mL-solution that consists of 9 mL of ropivacaine HCl 0.5% and 1 mL of dexamethasone 4mg/mL preparation) and injectate C (a total 25 mL solution that consists of 24 mL of ropivacaine HCl 0.5%, 1 mL of dexamethasone-4mg/mL preparation, and 0.125 mL of epinephrine-1:1000 preparation) at the end of procedure prior to the closure (which mimics standard care) is the control group
  Interventions: Drug: Normal Saline; Drug: Ropivacaine; Drug: Epinephrine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Normal Saline — Blocking the nerves between the ribs with a local anesthetic is normally done as a part of routine care at the end of the surgery in one set of injections. Intervention group will receive injectate A at the beginning and injectate B and C prior to the closure. Control group receive injectate B at the beginning of surgery and injectate A and C prior to the closure and end of surgery. Injectate B contains 10 mL of 0.9% normal saline.
Drug: Ropivacaine — Blocking the nerves between the ribs with a local anesthetic is normally done as a part of routine care at the end of the surgery in one set of injections. Intervention group will receive injectate A at the beginning and injectate B and C prior to the closure. Control group receive injectate B at the beginning of surgery and injectate A and C prior to the closure and end of surgery. Injectate A and C contain 9 and 24 mL of ropivacaine HCl 0.5%, respectively.
Drug: Epinephrine — Blocking the nerves between the ribs with a local anesthetic is normally done as a part of routine care at the end of the surgery in one set of injections. Intervention group will receive injectate A at the beginning and injectate B and C prior to the closure. Control group receive injectate B at the beginning of surgery and injectate A and C prior to the closure and end of surgery. Injectate C contains 0.125 mL of epinephrine-1:1000 preparation.
Drug: Dexamethasone — Blocking the nerves between the ribs with a local anesthetic is normally done as a part of routine care at the end of the surgery in one set of injections. Intervention group will receive injectate A at the beginning and injectate B and C prior to the closure. Control group receive injectate B at the beginning of surgery and injectate A and C prior to the closure and end of surgery. Injectates A and C both contain 1 mL of dexamethasone 4mg/mL preparation.

SUMMARY:
Intercostal nerve block, performed under the guidance of videoscope, is a part of standard anesthesia procedures for patients receiving Video-Assisted Thoracic Surgeries. In this double-blind, prospective, multi-center, randomized, controlled clinical trial the investigators aim to compare preemptive versus post-closure intercostal injection of ropivacaine in controlling post-video-assisted thoracotomy pain.

DETAILED DESCRIPTION:
The design of the study is a double-blind, prospective, multi-center, randomized, controlled clinical trial of preemptive vs. post-closure intercostal injection of ropivacaine in controlling post-video-assisted thoracotomy (VATS) pain. In standard intercostal nerve block procedures, the contents of A (a total of a 10 mL-solution that consists of 9 mL of ropivacaine HCl 0.5% and 1 mL of dexamethasone 4mg/mL preparation) and C (a total 25 mL solution that consists of 24 mL of ropivacaine HCl 0.5%, 1 mL of dexamethasone-4mg/mL preparation, and 0.125 mL of epinephrine-1:1000 preparation) are combined into one set of injections injected into the intercostal spaces of T5-6, T6-7, T7-8, T8-9 and T9-10, with each intercostal spaces receives about 7 mL of combined A and C solutions (each intercostal space receives 2 mL of A and about 5 mL of C). In this study, the intercostal nerve block is split into two sets of injections: one set of injections at the beginning of VATS, and the other set right before closure. Therefore the investigators consider both sets of injections as research procedures. Patients will be randomly assigned to receive a preemptive 2mL-injection of A or injection of B (contains 10 mL of 0.9% normal saline) at each intercostal space as previously delineated by the operating surgeon. Both the research team and the surgical team will be blind to the nature of the injectates during surgery. As parts of the standard care procedures, all patients will be monitored with non-invasive ASA standard in addition to invasive arterial blood pressure monitoring. Prior to the closure, patients who receive injections of A at the beginning of surgery will receive the second set of injections containing a mixture of B and C (5 mL of solution C is given at each intercostal space) at the intercostal spaces as previously delineated. Patients who receive injections of B at the beginning of surgery will receive the second set of injections containing a mixture of A and C (5 mL of solution C is given at each intercostal space). The investigators will group the patients who are assigned to receive injectate A at the end of the surgery as the control group. Because the injectate A and injectate C are usually given together in one set of injections at the same anatomical locations in standard intercostal nerve block procedures, the intercostal block received by the control group will closely resemble the procedures performed in standard intercostal nerve block. Patients who receive injectate A at the beginning of surgery are grouped as experimental group. Regardless of the group assignment, the total dosage of ropivacaine and dexamethasone given to a patient will be equal to the dosage given under the standard care procedures. Post operative pain, ventilatory profile and length of hospital stay will be compared between two study arms.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to enroll in this study if they:

* Have physical status within ASA class II or III
* Are between 18 and 85 years of age
* Are candidates for VATS
* Are able to complete VAS assessments
* Are competent to sign the informed consent form

Exclusion Criteria:

Patients will not be enrolled in this study if they:

* Are pregnant
* Have allergy to ropivacaine or hydromorphone
* Have renal insufficiency (eGFR<60mL/min/1.73m2)
* Have hepatic insufficiency (AST, ALT, or both >60 U/L) or cirrhosis
* Have a predicted postoperative forced vital capacity (FVC) of <40%, predicted forced expiratory volume at 1s (FEV1) <40%
* Have coagulopathy (platelet count<50000, INR>2, or both)
* Have a history of opioid addiction, chronically taking opioids, currently taking high dose of opioids or currently taking opioid agonist+antagonist (e.g. Suboxone®)
* Are taking nonsteroidal anti-inflammatory drug, including aspirin, within a week prior to surgery (since the analgesic effects of NSAID drugs may become confounding factors).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 0
  VAS scores at rest will be recorded right after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 6 hours
  VAS scores at rest will be recorded 6 hours after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 12 hours
  VAS scores at rest will be recorded 12 hours after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 18 hours
  VAS scores at rest will be recorded 18 hours after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 24 hours
  VAS scores at rest will be recorded 24 hours after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 48 hours
  VAS scores at rest will be recorded 48 hours after surgery and compared in both groups
Efficacy of intercostal nerve block in reducing postoperative pain, when performed at the beginning of video-assisted thoracic surgeries by visual analog scale (VAS) score | 72 hours
  VAS scores at rest will be recorded 72 hours after surgery and compared in both groups

SECONDARY OUTCOMES:
Postoperative delirium profiles measured using Intensive Care Delirium Screening Checklist (ICDSC) | 12 hours
  Postoperative delirium profiles will be measured 12 hours after surgery using Intensive Care Delirium Screening Checklist (ICDSC)
Postoperative delirium profiles measured using Intensive Care Delirium Screening Checklist (ICDSC) | 24 hours
  Postoperative delirium profiles will be measured 24 hours after surgery using Intensive Care Delirium Screening Checklist (ICDSC)
Postoperative delirium profiles measured using Intensive Care Delirium Screening Checklist (ICDSC) | 36 hours
  Postoperative delirium profiles will be measured 36 hours after surgery using Intensive Care Delirium Screening Checklist (ICDSC)
Postoperative delirium profiles measured using Intensive Care Delirium Screening Checklist (ICDSC) | 48 hours
  Postoperative delirium profiles will be measured 48 hours after surgery using Intensive Care Delirium Screening Checklist (ICDSC)
PaO2/FIO2 ratio right after surgery | 0 hours
  PaO2 (mmHg kPa) and FIO2 (percent) will be recorded from atrial blood gas examination and the ratio will be calculated
Total hospital length of stay | up to 2 weeks
  The investigators will assess length of stay by evaluating medical records and calculate length of stay in days, using date of discharge and date of admission
Need for non-invasive positive pressure ventilation (NIPPV) | up to two weeks
  The investigators will assess the need for NIPPV by evaluating medical records to asses if patients received NIPPV with the discretion of the managing physician during their hospitalization
Need for mechanical ventilation | up to two weeks
  The investigators will assess the need for mechanical ventilation by evaluating medical records to asses if patients received mechanical ventilation with the discretion of the managing physician during their hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- VA Western New York Healthcare System, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
The investigators don't plan to make individual participant data (IPD) available to other researchers.